CLINICAL TRIAL: NCT02415881
Title: Phase I, Open-label Study Evaluating the Safety and Pharmacokinetics of Escalating Doses of Panitumumab-IRDye800 as an Optical Imaging Agent to Detect Head and Neck Cancer During Surgical Procedures
Brief Title: Panitumumab IRDye800 Optical Imaging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eben Rosenthal (Other)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35064; ENT0050 (Other: OnCore)
Record Dates: First submitted 2015-03-26; First posted 2015-04-14 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer
Keywords: Panitumumab; Optical Imaging
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Panitumumab IRDye 800 (Experimental): Patients will receive Panitumumab IRDye800 prior to their scheduled surgery.
  Interventions: Drug: Panitumumab IRDye 800; Device: da Vinci Firefly; Device: IMAGE1 + ICG Hopkins telescope and/or VITOM

INTERVENTIONS:
Drug: Panitumumab IRDye 800 — Patients will receive Panitumumab IRDye 800 prior to their scheduled surgery
  Other Names: Optical Imaging prior to surgery
Device: da Vinci Firefly — Da Vinci surgical robot with build-in fluorescence imaging option (Firefly technology)
Device: IMAGE1 + ICG Hopkins telescope and/or VITOM — IMAGE1 + ICG Hopkins telescope and/or VITOM -- Fluorescence camera allowing for imaging of IRDye800. Camera is suitable for open and laparoscopic surgery.

SUMMARY:
Phase I trial to evaluate the safety of escalating dose levels of conjugated panitumumab-IRDye800 in subjects with head and neck squamous cell carcinoma (HNSCC) that undergo surgery with curative intent.

DETAILED DESCRIPTION:
This is a Phase I trial that is designed to evaluate the safety of escalating dose levels of conjugated panitumumab-IRDye800 used in subjects with head and neck squamous cell carcinoma (HNSCC) that undergo surgery with curative intent. Safety data from this trial will be studied to assist in the selection of dose levels of panitumumab-IRDye800 for future research. It is hoped that this study will also help in finding better methods for identifying cancer intraoperatively for a more complete surgical resection.

ELIGIBILITY:
Inclusion Criteria

* Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck
* Patients diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Patients with recurrent disease or a new primary will be allowed.
* Planned standard of care surgery with curative intent for squamous cell carcinoma
* Age ≥ 19 years
* Have life expectancy of more than 12 weeks
* Karnofsky performance status of at least 70% or ECOG/Zubrod level 1
* Have acceptable hematologic status, coagulation status, kidney function, and liver function including the following clinical results: Hemoglobin ≥ 9 gm/dL; White blood cell count > 3000/mm3; Platelet count ≥ 100,000/mm3; Serum creatinine ≤ 1.5 times upper reference range

Exclusion Criteria

* Received an investigational drug within 30 days prior to first dose of panitumumab IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions monoclonal antibody therapies
* Pregnant or breastfeeding
* Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females)
* Magnesium or potassium lower than the normal institutional values
* Patients receiving Class IA (quinidine, procanamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Patients with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* TSH > 13 micro International Units/mL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Safety profile of panitumumab conjugated panitumumab IRDye800 will be measured by assessing number of Grade 2 or higher adverse events | 30 days
  Safety profile of panitumumab conjugated to IRDye800CW (panitumumab IRDye800) will be measured by assessing number of Grade 2 or higher adverse events which have been determined to be clinically significant and definitely, probably or possibly related.

SECONDARY OUTCOMES:
Efficacy of panitumumab IRDye800 will be measured by tumor to background ratio | 7 days
  Efficacy of panitumumab IRDye800 will be measured by tumor to background ratio. Fluorescence intensity of tumor tissue compared to that of normal surrounding tissue.
Optimal timing of the surgical procedure to maximize tumor to background ratio | 7 days
  Fluorescence intensity of tissue obtained from patients undergoing surgery at different time points in various cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Eben L Rosenthal, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Stanford University, School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu G, Nishio N, van den Berg NS, Martin BA, Fakurnejad S, van Keulen S, Colevas AD, Thurber GM, Rosenthal EL. Co-administered antibody improves penetration of antibody-dye conjugate into human cancers with implications for antibody-drug conjugates. Nat Commun. 2020 Nov 9;11(1):5667. doi: 10.1038/s41467-020-19498-y. PMID 33168818
- [Derived] Kapoor S, Lu G, van den Berg NS, Krishnan G, Pei J, Zhou Q, Martin BA, Baik FM, Rosenthal EL, Nishio N. Effect of Formalin Fixation for Near-Infrared Fluorescence Imaging with an Antibody-Dye Conjugate in Head and Neck Cancer Patients. Mol Imaging Biol. 2021 Apr;23(2):270-276. doi: 10.1007/s11307-020-01553-1. Epub 2020 Oct 19. PMID 33078373
- [Derived] Fakurnejad S, van Keulen S, Nishio N, Engelen M, van den Berg NS, Lu G, Birkeland A, Baik F, Colevas AD, Rosenthal EL, Martin BA. Fluorescence molecular imaging for identification of high-grade dysplasia in patients with head and neck cancer. Oral Oncol. 2019 Oct;97:50-55. doi: 10.1016/j.oraloncology.2019.08.008. Epub 2019 Aug 12. PMID 31421471